CLINICAL TRIAL: NCT06862804
Title: The Effect of Applied Group Training Given to Mothers With Children With Autism on Perceived Social Support, Depressive Symptoms and Self-compassion: A Randomised Controlled Trial
Brief Title: The Effect of Applied Group Training Given to Mothers With Children With Autism on Perceived Social Support, Depressive Symptoms and Self-compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Havva Kaçan, ASSOCIATE PROFESSOR, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-KAEK-117; 2024-KAEK-117 (Other: Kastamonu University)
Record Dates: First submitted 2025-02-14; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Parent
Keywords: parents; special needs child; self-compassion; perceived social support; depressive symptoms; autism; autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The data obtained in the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 programme. Number, percentage, mean, standard deviation will be used as descriptive statistical methods in the evaluation of the data. The homogeneity of the descriptive characteristics according to the groups will be analysed by chi-square and t-test. The kurtosis and skewness values related to the normal distribution of the scale scores will be examined and the reference value ranges (+2.0 and -2.0; George, & Mallery, 2010) will be determined, the difference of the scale scores between the groups will be analysed by independent samples t-test and the change within the group will be analysed by dependent samples t-test (paired samples). Cronbach's alpha values will be calculated when calculating the reliability coefficients of the scales. For all statistical analyses, the significance level will be accepted as p<0.05.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Those receiving group training (Experimental): TThe group training programme will be completed in six consecutive weeks, two per week, and the caregivers will be divided into two groups of 12 people with the support of the school administration according to their attendance at the school. The first group will be organised on Tuesday and the second group on Friday. For those who cannot attend both groups, weekly training will be given on Saturdays. Each group session will last 45-60 minutes, the first 10 minutes will be spent summarising the previous session, 40 minutes will be spent implementing the plan in line with the session topic, the last 10 minutes will be spent evaluating and summarising the session and ending the session by explaining the next session topic.
  No application will be made to the individuals in the control group during the study. The pretest scales will be applied individually by the researchers when the participants come to the unit to give information about the study and to obtain voluntary consent.
  Interventions: Behavioral: practical group training
- those who do not receive group training (Active Comparator): no intervetion
  Interventions: Behavioral: practical group training

INTERVENTIONS:
Behavioral: practical group training — It is understood how important the issue is when it is considered that supporting these families, especially mothers, both socially and psychologically can be important in alleviating the difficulties they experience and that mothers with children with autism are in a risk group in terms of receiving this support. The research was designed considering that the applied training we will provide will be effective in increasing social support and developing self-compassion for the primary caregivers of children and will reduce the level of depressive symptoms.
  Arms: Those receiving group training
Behavioral: practical group training — practical group training
  Arms: those who do not receive group training

SUMMARY:
Autism Spectrum Disorder (ASD), which can also be defined as a type of special need, is a congenital neurodevelopmental disorder whose symptoms are observed in early childhood. ASD, which has deficits in social communication and interaction as well as limited-repetitive behaviour patterns, starts in the early developmental stage and causes a significant impairment in areas of social functioning .

A child with autism causes serious anxiety and depression in the family for many reasons, including the uncertainty of the diagnosis, the severity and duration of the disorder, and the child's lack of compliance with social rules. ASD has devastating effects not only on the individual but also on carers . It is reported that mothers with a child with ASD experience psycho-social difficulties compared to parents with a normally developing child . Hyperactivity, mood problems, disturbances in sleep and eating patterns, obsessions and compulsive behaviours, and self-injurious behaviours of children with ASD make the parent-child relationship difficult. Due to the burden of care brought about by such findings and difficulties, the family begins to experience situations such as decreased quality of relationship between family members, educational problems, financial difficulties and future anxiety. There is a significant relationship between emotional and behavioural problems of children with ASD and anxiety and depression levels of their parents.

In addition to psychological symptoms, caregiver parents also experience limitations in daily life activities. The ability of mothers with children with autism to cope with unexpected situations is closely related to the social support they perceive. However, studies show that parents with children with autism have difficulties in entering and adapting to the society, and therefore, friends, neighbours and close environment relations from which they can get social support are weakened. Considering that supporting these families, especially mothers, both socially and spiritually can be important in alleviating the difficulties they experience and that mothers with autistic children are in a risk group in terms of receiving this support, it is understood how important the issue is.

Self-compassion is the individual's directing compassionate behaviours and attitudes towards himself/herself. Neff defines self-compassion as individuals being kind and compassionate towards themselves in difficult situations of inadequacy, failure and pain, accepting their negative emotions by being aware of them, and knowing that all kinds of challenging situations that can be experienced are related to being human. Self-compassion is recognised as one of the healthy ways of coping with difficult experiences and pain. It is stated that self-compassion is positively associated with coping strategies such as active coping, acceptance and reorganisation, and negatively associated with coping strategies such as mental-behavioural dissolution or rejection. In the findings of self-compassion-based studies conducted with parents who have children with disabilities in the literature, it was reported that as the level of self-compassion increases, parents' optimism levels increase, self-compassion has a negative relationship with burnout and a positive relationship with subjective well-being, and positive coping strategies increase as the level of self-compassion increases.

H0: The applied training programme has no effect on perceived social support, depressive symptoms and self-compassion.

H1: The applied training programme has an effect on perceived social support, depressive symptoms and self-compassion.

Sample of the research:The population of the study consists of caregivers who have children between the ages of 6-18 years with autism diagnosed with autism who are educated in 3 special education and rehabilitation centres in Kastamonu province and who undertake their primary care. Caregivers who brought their children to these centres for the purpose of education, who meet the research criteria and who voluntarily accept to participate in the research will be included in the sample. Power analysis was performed with the G*Power 3.1 programme to determine the number of people to be included in the sample, and it was planned to include 48 caregivers, 24 in the experimental group and 24 in the control group.

DETAILED DESCRIPTION:
* Data Collection Tool: Data collection tools consist of four parts.

  1. Descriptive characteristics form: It consists of eight questions about the descriptive characteristics of the child with autism and the caregiver, including questions about the caregiver's age, gender, education level, and problems encountered in care.
  2. Multidimensional Perceived Social Support Scale: The original form was developed by Zimet et al. (1988) in the United States of America and its adaptation to Turkish, reliability and validity study was conducted by Eker, Arkar, Yaldız (2001). With the Multidimensional Perceived Social Support Scale, the adequacy of social support received from three different sources is subjectively evaluated. The Likert-type scale, which is scored from 1 to 7, ranges from 4 to 28 for the sub-dimensions and from 12 to 84 for the total score of the scale. A high score indicates that the perceived social support is high.
  3. Beck Depression Inventory: It was developed in 1978 by Beck et al. to measure depression levels of individuals. Beck Depression Inventory is a frequently used inventory that measures emotional, physical, cognitive and motivational symptoms of depression. The purpose of the Beck Depression Inventory is not to diagnose but to objectively measure the depression level of the individual. Its Turkish validity and reliability was carried out by Durak and Palabıyıkoğlu in 1994. Each of the subcategories in the scale consists of 4 items and is graded with 0 to 3 points. A maximum score of 63 and a minimum score of 0 can be obtained. Scores between 0-9 points are considered as normal, 16-23 as moderate depression, 24-63 as severe depression.
  4. Self-Compassion Scale:

     It is a self-report scale developed by Neff (2003) and adapted to Turkish by Akın et al. (2007). It consists of a total of 6 sub-dimensions and 26 items: Self-Compassion, Self-Judgement, Awareness of Sharing, Isolation, Consciousness and Overidentification. The score of the 5-point Likert-type scale varies between 26 and 130. Since selfjudgement, isolation and overidentification are negative subscales, their items are reverse coded. The averages of the six subscales give the total mean of self-compassion. Mean scores between 1-2.5 indicate low level of self-compassion, scores between 2.5-3.5 indicate medium level of self-compassion and scores between 3.5-5 indicate high level of self-compassion. The internal consistency coefficients of the scale were found between .72 and .80.

     Data Collection Process

     The data will be collected face-to-face by the researchers when the caregivers bring their children to their institutions. In the preliminary preparation phase; the author (HK) will inform the unit managers of the centres where the study will be conducted about the aims of the study and the application processes, the personal data form and scales will be applied by the researcher in a quiet classroom environment, after the individuals to be included in the experimental and control groups are determined, the preliminary data will be collected from both groups before the training is given. The group training programme will be completed in six consecutive weeks, two per week, and the caregivers will be divided into two groups of 12 people with the support of the school administration according to their arrival to the school. The first group will be organised on Tuesday and the second group on Friday. For those who cannot attend both groups, weekly training will be given on Saturdays. Each group session will last 45-60 minutes, the first 10 minutes will be spent summarising the previous session, 40 minutes will be spent implementing the plan in line with the session topic, the last 10 minutes will be spent evaluating and summarising the session and ending the session by explaining the next session topic.

     No application will be made to the individuals in the control group during the study. The pretest scales will be applied individually by the researchers when the participants come to the unit to give information about the study and to obtain voluntary consent. The post-test will be administered six weeks after the pre-test at the same place and by the same researchers.

     Sessions

  <!-- -->

  1. Meeting with the group members, introduction of the group process, explanation of the session topics,
  2. Difficulties in caring for a child with autism and coping behaviours
  3. Self-Compassionate approach training practices
  4. I discover my strengths through painting activities for the recognition and expression of emotions.
  5. Gaining Positive Health Behaviours: Interpersonal communication and using supports, anger management
  6. Gaining Positive Health Behaviours: Managing Stress, Progressive relaxation techniques and taking questions
* Data Analysis:

The data obtained in the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 programme. Number, percentage, mean, standard deviation will be used as descriptive statistical methods in the evaluation of the data. The homogeneity of the descriptive characteristics according to the groups will be analysed by chi-square and t-test. The kurtosis and skewness values related to the normal distribution of the scale scores will be examined and the reference value ranges (+2.0 and -2.0; George, & Mallery, 2010) will be determined, the difference of the scale scores between the groups will be analysed by independent samples t-test and the change within the group will be analysed by dependent samples t-test (paired samples). Cronbach's alpha values will be calculated when calculating the reliability coefficients of the scales. For all statistical analyses, the significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Being a parent of a child diagnosed with autism spectrum disorder between the ages of 1-18
2. To have assumed the responsibility of giving primary care to the child with autism,
3. Having provided care for at least 6 months,

Exclusion Criteria:

* 1-Mental or physical disability, 2-Having participated in a similar training programme before

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women
Enrollment: 44 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
The effect of the implemented training program on Perceived Social Support will be measured. | Four Week
  The effect of the implemented training program on Perceived Social Support and its level will be measured with the Perceived Social Support scale.

SECONDARY OUTCOMES:
The psychosocial status assessment level of parents will be measured with the Psychosocial Status Assessment Scale for Parents (1-3 years). | Four Week
  The psychosocial status assessment level of parents will be measured with the Psychosocial Status Assessment Scale for Parents (1-3 years).

OTHER OUTCOMES:
The severity of depressive symptoms will be measured with the Beck Depression Inventory for the effect of applied group training given to mothers of children with autism on depressive symptoms. | four week
  The severity of depressive symptoms will be measured with the Beck Depression Inventory for the effect of applied group training given to mothers of children with autism on depressive symptoms.
The self-compassion level of parents of autistic children will be measured with the self-compassion scale. | Four Week
  The self-compassion level of parents of autistic children will be measured with the self-compassion scale.

CONTACTS AND LOCATIONS:
Overall Officials: Havva KAÇAN, ASSOCIATE PROFESSOR DOCTOR, Principal Investigator — Kastamonu University; Şevval YEYİT, Research Assistant, Study Chair — Kastamonu University; Vasfiye Bayram Değer, ASSOCIATE PROFESSOR DOCTOR, Study Chair — Mardin Artuklu University
Locations (1):
- Kastamonu private educational institutions, Kastamonu, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided